CLINICAL TRIAL: NCT05018637
Title: Efficacy of Wharton's Jelly-derived Mesenchymal Stem Cells in Combination With Parathyroid Hormone for Vertebral Compression Fracture
Brief Title: Efficacy of WJ-derived Mesenchymal Stem Cells in Combination With Parathyroid Hormone for Vertebral Compression Fracture
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Inbo Han (Other)
Responsible Party: Sponsor-Investigator, Inbo Han, Principal Investigator, Professor of Spine neurosurgeon, MD, PhD, CHA University
Organization: CHA University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-11-010
Record Dates: First submitted 2021-08-15; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Vertebral Compression Fracture; Osteoporotic Fractures
Keywords: vertebral compression fracture; Back Pain
MeSH Terms: conditions — Osteoporotic Fractures; Back Pain | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WJ-MSC group (Experimental): intramedullary injection of 4 x 107 WJ-MSCs (direct injection into the recently fractured vertebra) at baseline (day 0). subcutaneous injection of 20 µg teriparatide once daily for 6 months, followed by oral administration of anti-resorptive drug for 6 months.
  Interventions: Drug: WJ-MSC; Drug: Teriparatide
- Teriparatide group (Active Comparator): subcutaneous injection of 20 µg teriparatide once daily for 6 months, followed by oral administration of anti-resorptive drug for 6 months.
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: WJ-MSC — Other: subcutaneous injection of 20 µg teriparatide once daily for 6 months, followed by oral administration of anti-resorptive drug for 6 months.
  Other: intramedullary injection of 4 x 107 WJ-MSCs (direct injection into the recently fractured vertebra) at baseline (day 0). subcutaneous injection of 20 µg teriparatide once daily for 6 months, followed by oral administration of anti-resorptive drug for 6 months.
  Other Names: teriparatide
  Arms: WJ-MSC group
Drug: Teriparatide — subcutaneous injection of 20 µg teriparatide once daily for 6 months, followed by oral administration of anti-resorptive drug for 6 months.

SUMMARY:
Osteoporotic vertebral compression fractures (OVCFs) are serious health problems. Transplantation of mesenchymal stem cells (MSCs) has gained considerable attention to treat osteoporosis and OVCFs because implanted healthy MSCs could be differentiated into osteoblasts and reduce the susceptibility of fractures by facilitating new bone formation.

This study compares teriparatide (PTH 1-34) injection to combined treatment with Wharton's jelly-derived MSCs (WJ-MSCs) and teriparatide (PTH 1-34) in patients with OVCFs.

It is a randomized, open-label, phase 2 study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women over 40 years of age
* Compression fracture of the spine confirmed by MRI or bone scan

  * When the T score of the lumbar spine is less than -1.0 in the bone density test using DXA (Dual energy X ray absorptiometry)
  * Compression fracture is between 5th thoracic and 5th lumbar vertebra
  * When a new vertebral fracture occurs in less than 3 parts of the spine
  * Compression fracture of the spine within 6 weeks after minor trauma
* Oswestry Disability Index (ODI) due to vertebral fracture is more than 30%
* Back pain due to vertebral fracture has a Visual Analogue Scale (VAS) of 4 or higher.
* In case of writing consent for stem cell transplantation therapy

Exclusion Criteria:

* Those who used osteoporosis treatment (bisphosphonate, selective estrogen receptor modulator, or parathyroid hormone) 6 months before the start of the clinical trial due to osteoporotic vertebral fracture.
* In the case of inherited, metabolic, neoplastic, or infectious bone disease other than osteoporosis
* Spinal fracture with neurological symptoms
* Those who are taking drugs that affect bone metabolism such as steroids.
* Those who have undergone spinal fixation surgery on the fracture site prior to the clinical trial
* Those who have a history of psychiatry or who are currently undergoing treatment, who have judged that it is difficult to proceed with the clinical trial under the judgment of the researcher
* Those who do not understand the purpose and method of this clinical trial as a study subject for drug or alcohol addiction
* Those who participated in other clinical trials within 30 days prior to participation in the clinical trial
* Those who may affect this clinical trial due to serious medical conditions (hypertension not controlled by drugs, diabetes not controlled by drugs, blood coagulation disease, cirrhosis, kidney failure, tumor) or immune deficiency
* Factors less than 10 g/dL of hemoglobin in general blood test
* If there is currently an acute systemic or local infection
* Others who have clinically significant findings deemed inappropriate for this clinical trial due to medical judgment by the person in charge of the clinical trial
* Those who are allergic to proteins required for cell production (fetal calf serum)

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
improvement in Visual Analogue Scale | 12 months
  Change in the VAS at 1, 3, 6, 9, and 12 months after the transplantation of Wharton's jelly-derived MSCs (WJ-MSCs), compared to before the transplantation.
  on a scale of 0 to 10, with 0 meaning no pain and 10 meaning the worst pain you can imagine.

SECONDARY OUTCOMES:
improvement in Oswestry Disability Index | 12 months
  Change in the ODI at 1, 3, 6, 9, and 12 months after the transplantation of WJ-MSCs, compared to before the transplantation.
  on a scale of 0 to 3, with 0 meaning no disability and 10 meaning severe disability
Change in the T score (lumbar spine and femoral neck) of dual-energy x-ray absorptiometry | 12 months
  Change in the T score (lumbar spine and femoral neck) of dual-energy x-ray absorptiometry at 6 and 12 months after the transplantation compared to before the transplantation
Presence of new vertebral fracture | 12 months
  identification of spine fracture based on x ray
Change in the bone mineral density (computed tomography) of fractured vertebrae | 12 months
  Change in the bone mineral density (computed tomography) at 6 and 12 months after the transplantation compared to before the transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- CHA University, CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea